CLINICAL TRIAL: NCT00889473
Title: A Phase IIb, Randomized, Double-blind, Placebo Controlled, Dose Ranging, Multicenter Study to Determine the Safety, Tolerance, and Efficacy of Larazotide Acetate (AT-1001) in Celiac Disease Subjects During a Gluten Challenge
Brief Title: Study of the Efficacy of Larazotide Acetate to Treat Celiac Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: 9 Meters Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLIN1001-006 Part B
Record Dates: First submitted 2009-04-27; First posted 2009-04-29 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Celiac Disease
Keywords: larazotide acetate; gluten
MeSH Terms: conditions — Celiac Disease | interventions — larazotide acetate; Glutens

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo-controlled, dose ranging, multicenter
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Larazotide acetate 1 mg (Experimental): larazotide acetate 1 mg capsules TID + 900 mg gluten capsules TID for 6 weeks
  Interventions: Drug: Larazotide acetate; Dietary Supplement: Gluten 900 mg
- Placebo (Placebo Comparator): placebo capsules TID + 900 mg gluten capsules TID for 6 weeks
  Interventions: Drug: Placebo; Dietary Supplement: Gluten 900 mg

INTERVENTIONS:
Drug: Larazotide acetate — gelatin capsule
  Other Names: AT1001; INN-202
  Arms: Larazotide acetate 1 mg
Drug: Placebo — gelatin capsule
  Arms: Placebo
Dietary Supplement: Gluten 900 mg — gelatin capsule

SUMMARY:
This study is designed to evaluate the efficacy of a single dose of larazotide acetate in preventing intestinal permeability changes induced by a 6-week gluten challenge in subjects with celiac disease

DETAILED DESCRIPTION:
This study is an extension of Study CLIN1001-006 (NCT 00492960). This is a Phase IIb, randomized, double-blind, placebo-controlled, dose ranging, multicenter study to determine the safety, tolerance, and efficacy of larazotide acetate in subjects with celiac disease during a gluten challenge. Subjects will remain on their gluten-free diet throughout the duration of the trial.

Study drug or drug placebo capsules will be administered TID 15 minutes before each meal. Gluten or gluten placebo capsules will be taken TID with each meal.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults with biopsy proven celiac disease on a gluten-free diet for at least the past 6 months
* Anti-Tissue Transglutaminase (anti-tTG) ≤ 10 EU.
* BMI between 18.5 and 38, inclusive.

Exclusion Criteria

* Has chronic active GI disease other than celiac disease
* Has diabetes (Type 1 or Type 2).
* Unable to abstain from alcohol consumption or NSAID use for 48 hours prior to each intestinal permeability collection throughout the study.
* Has hemoglobin value below 8.5 g/dL

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-04 (Actual); Primary Completion 2009-11 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Response to gluten | 6 weeks

SECONDARY OUTCOMES:
Anti-transglutaminase | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Leon, MD, PhD, Study Director — Alba Therapeutics Inc
Locations (15):
- United States (14):
  - Study Site, Orange, California
  - Study Site, Topeka, Kansas
  - Study Site, Lexington, Kentucky
  - Study Site, Hagerstown, Maryland
  - Study Site, Silver Spring, Maryland
  - Study Site, Chesterfield, Michigan
  - Study Site, Troy, Michigan
  - Study Site, Rochester, Minnesota
  - Study Site, New York, New York
  - Study Site, Oklahoma City, Oklahoma
  - Study Site, Paoli, Pennsylvania
  - Study Site, Philadelphia, Pennsylvania
  - Study Site, Pittsburgh, Pennsylvania
  - Study Site, Franklin, Tennessee
- Study Site, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No